CLINICAL TRIAL: NCT04628767
Title: A Phase II/III Trial of Durvalumab and Chemotherapy for Patients With High Grade Upper Tract Urothelial Cancer Prior to Nephroureterectomy
Brief Title: Testing the Addition of MEDI4736 (Durvalumab) to Chemotherapy Before Surgery for Patients With High-Grade Upper Urinary Tract Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-09850; NCI-2020-09850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8192 (Other: ECOG-ACRIN Cancer Research Group); EA8192 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Renal Pelvis and Ureter Urothelial Carcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; durvalumab; Immunoglobulin G; Disulfides; Gemcitabine; Magnetic Resonance Spectroscopy; Methotrexate; merphos; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A (durvalumab, chemotherapy) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 of chemotherapy cycles 1 and 3. Patients also receive methotrexate IV over 2-3 minutes, vinblastine sulfate IV, doxorubicin IV, cisplatin IV over at least 2 hours on day 1. Treatments repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 21- 60 days after completion of systemic treatment, patients with continued lack of radiographic presence of metastatic or unresectable disease undergo surgery. Patients also undergo tissue biopsy and blood sample collection on study, and CT or MRI throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Biological: Pegfilgrastim; Procedure: Therapeutic Conventional Surgery; Drug: Vinblastine Sulfate
- Arm B (chemotherapy) (Active Comparator): Patients also receive methotrexate IV over 2-3 minutes, vinblastine sulfate IV, doxorubicin IV, cisplatin IV over at least 2 hours on day 1. Treatments repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 21- 60 days after completion of systemic treatment, patients with continued lack of radiographic presence of metastatic or unresectable disease undergo surgery. Patients also undergo tissue biopsy and blood sample collection on study, and CT or MRI throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Biological: Pegfilgrastim; Procedure: Therapeutic Conventional Surgery; Drug: Vinblastine Sulfate
- Arm C (durvalumab, gemcitabine hydrochloride) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 21- 60 days after completion of systemic treatment, patients with continued lack of radiographic presence of metastatic or unresectable disease undergo surgery. Patients also undergo tissue biopsy and blood sample collection on study, and CT or MRI throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm A (durvalumab, chemotherapy); Arm B (chemotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Doxorubicin Hydrochloride — Given Iv
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Arm A (durvalumab, chemotherapy); Arm B (chemotherapy)
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Arm A (durvalumab, chemotherapy); Arm C (durvalumab, gemcitabine hydrochloride)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Arm C (durvalumab, gemcitabine hydrochloride)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm A (durvalumab, chemotherapy); Arm B (chemotherapy)
Biological: Pegfilgrastim — Given via injection
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
  Arms: Arm A (durvalumab, chemotherapy); Arm B (chemotherapy)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: Vinblastine Sulfate — Given Iv
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE
  Arms: Arm A (durvalumab, chemotherapy); Arm B (chemotherapy)

SUMMARY:
This phase II/III trial compares the effect of adding durvalumab to chemotherapy versus chemotherapy alone before surgery in treating patients with upper urinary tract cancer. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as methotrexate, vinblastine, doxorubicin, cisplatin, and gemcitabine work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Durvalumab in combination with chemotherapy before surgery may enhance the shrinking of the tumor compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare event-free survival (EFS) between patients with upper tract urothelial cancer (UTUC) randomized to neoadjuvant accelerated methotrexate, vinblastine, adriamycin, cisplatin (aMVAC) alone or in combination with durvalumab. (Cisplatin eligible patients [Arms A and B]) II. Evaluation of pathologic complete response at radical nephroureterectomy (RNU) (pathologic complete response [pCR], ypT0N0/ Nx). (Cisplatin ineligible patients [Arm C]).

SECONDARY OBJECTIVES:

I. To assess pathologic complete response (pCR) at surgery. (Cisplatin eligible cohort) II. Event-free survival (EFS) will be evaluated for the cisplatin ineligible cohort as a secondary endpoint. (Cisplatin ineligible cohort) III. Overall survival in all, and by post chemotherapy response (ypt0N0, yp =< T1N0, yp >= T2Nany). (All patients) IV. To evaluate disease-free survival (DFS) in each arm of the trial separately. (All patients) V. To evaluate cancer-specific survival of patients in each arm of the trial separately. (All patients) VI. To evaluate renal function outcomes following systemic treatment and following surgery ([RNU) in each arm of the trial separately. (All patients) VII. To evaluate safety and tolerability of neoadjuvant aMVAC alone or in combination with durvalumab prior to RNU. (All patients)

OUTLINE: Patients eligible for cisplatin are randomized to Arms A or B. Patients ineligible for cisplatin are assigned to Arm C.

ARM A: Patients receive durvalumab intravenously (IV) over 60 minutes on day 1 of chemotherapy cycles 1 and 3. Patients also receive methotrexate IV over 2-3 minutes, vinblastine sulfate IV, doxorubicin IV, cisplatin IV over at least 2 hours on day 1. Treatments repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 21- 60 days after completion of systemic treatment, patients with continued lack of radiographic presence of metastatic or unresectable disease undergo surgery.

ARM B: Patients also receive methotrexate IV over 2-3 minutes, vinblastine sulfate IV, doxorubicin IV, cisplatin IV over at least 2 hours on day 1. Treatments repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 21- 60 days after completion of systemic treatment, patients with continued lack of radiographic presence of metastatic or unresectable disease undergo surgery.

ARM C: Patients receive durvalumab IV over 60 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 21- 60 days after completion of systemic treatment patients with continued lack of radiographic presence of metastatic or unresectable disease undergo surgery.

Patients also undergo tissue biopsy and blood sample collection on study, and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up within 30 days and then every 3-6 months for up to 5 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION AND RANDOMIZATION
* Patients must be >= 18 years of age
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Patient must have a diagnosis of high grade upper tract urothelial carcinoma expected within 14 weeks (98 days) prior to registration/randomization with one of the following:

  * Biopsy (gold standard, preferred) and either upper urinary tract mass on cross-sectional imaging or
  * Tumor directly visualized during upper urinary tract endoscopy
  * High grade cytology and clinically estimated invasive upper urinary tract mass on cross-sectional imaging (e.g., including presence of tumor-related hydronephrosis) or tumor directly visualized during upper urinary tract endoscopy

    * NOTE: Universal histologic testing of UTUC with additional studies, such as immunohistochemistry or microsatellite instability, is strongly recommended to identify patients with high probability of Lynch-related or other germline mutation related cancers whom clinicians should refer for genetic counseling and germline testing (this is not required for eligibility)

      * Due to the anatomy of upper urinary tract and lack of muscularis propria, pathologic evidence of cT2 on biopsy is usually not possible
* Leukocytes >= 3,000/mcL (obtained =< 14 days prior to registration/randomization)
* Platelets >= 100,000/mcL (obtained =< 14 days prior to registration/randomization)
* Total bilirubin =< 1.2 mg/dL (or ≤ 2 mg/dLfor patients with Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x institutional ULN (obtained =< 14 days prior to registration/randomization)
* Hemoglobin (Hgb) >= 9 g/dL (obtained =< 14 days prior to registration/randomization)

  * NOTE: Packed red blood transfusion is allowed to achieve this parameter as per treating investigator
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration/randomization are eligible for this trial

  * NOTE: These patients must be stable on their anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on the same regimen; the most recent undetectable viral load must be within the past 12 weeks. They must have a CD4 count of greater than 250 cells/mcL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/mcL over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy induced bone marrow suppression. They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months
  * NOTE: For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/mcL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy. They must have an undetectable viral load and a CD4 count >= 250 cells/mcL within 7 days of registration/randomization
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * NOTE: Testing for HIV, hepatitis B or hepatitis C is not required unless clinically indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and have undetectable viral load. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patient must have a body weight of > 30 kg
* Patient must have life expectancy of >= 12 weeks
* Patient must have creatinine clearance > 15 ml/min as estimated by Cockcroft-Gault formula or glomerular filtration rate (GFR) > 15 ml/min/1.73m^2 within 28 days prior to registration/randomization

  * NOTE: Patients will be assigned to cisplatin-ineligible and cisplatin-eligible cohorts based on their creatinine clearance, Eastern Cooperative Oncology Group (ECOG) performance status, and grade (if any) of peripheral neuropathy and/or hearing loss in keeping with recommended cisplatin contraindications. Patients who are cisplatin-eligible will be randomized to either Arm A or Arm B and patients who are cisplatin-ineligible will be registered to Arm C

    * Patients that meet any of the following four criteria will be registered to the cisplatin-ineligible Arm C if they meet other eligibility criteria:

      * Creatinine clearance > 15 ml/min and =< 50 ml/min (estimated by Cockcroft-Gault formula) or GFR > 15ml/min/1.73m^2 and ≤ 50 ml/min/1.73 m^2
      * Hearing loss >= 3
      * Neuropathy >= 2
      * ECOG performance status 2
    * In addition, the patient must have an absolute neutrophil count (ANC) >= 1,000/mcL obtained =< 14 days prior to registration
    * Patients that meet all of the following four criteria will be randomized to the cisplatin-eligible Arm A or Arm B:

      * Creatinine clearance of > 50ml/min (estimated by Cockcroft-Gault formula) or GFR > 50ml/min/1.73m^2
      * ECOG performance status 0-1
      * Hearing loss grade 0-2
      * Neuropathy 0-2
    * In addition, the patient must have an absolute neutrophil count (ANC) >= 1,500/mcL obtained =< 14 days prior to randomization
    * Also, the patient must have left ventricular ejection fraction (LVEF) >= 50% by (either multigated acquisition scan [MUGA] or 2-D echocardiogram) obtained within obtained within 28 days prior to randomization

Exclusion Criteria:

* Patients must not have any component of small cell/neuroendocrine carcinoma. Other histologic subtypes (variants) are permitted provided the half or predominant (>= 50%) subtype is conventional urothelial carcinoma
* Patients must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy. A patient of childbearing potential is defined as any patient, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients of childbearing potential and sexually active patients must not expect to conceive or father children, either by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse from the time of registration, while on study treatment and for at least 6 months after the last dose of protocol treatment
* Patients must have no evidence of metastatic disease or clinically enlarged regional lymph nodes (>= 1.5 cm short axis) on imaging required within 28 days prior to registration (Non-regional findings >=1.5 cm short axis that in the opinion of the investigator are not concerning for involvement based on radiographic characteristics, chronicity, avidity on positron emission tomography (PET) or other imaging or other criteria can be eligible based on investigator discretion).

  * NOTE: Patients with elevated alkaline phosphatase, calcium or suspicious bone pain/tenderness can also undergo baseline bone scan to evaluate for bone metastasis at the discretion of local provider.
* Patient must meet below criteria for prior/current malignancy history:

  * Non-urothelial cancer malignancy history:

    * Patient must not have another active (or within two years) second malignancy other than resected non-melanoma skin cancers, resected in situ breast, cervical or other in situ carcinoma, and either clinically insignificant per the investigator (e.g. =< Gleason 3+4) on active surveillance (or watchful waiting) or previously treated prostate cancer with no rising prostate specific antigen (PSA) and no plan to treat

      * NOTE: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
    * Urothelial cancer malignancy history:

      * Patient may have a history of resectable urothelial cancer as long as patients meet one of the following:
      * T0, Ta or Tis at any time
      * T1-4a N0 and no evidence of disease (NED) for more than 2 years from the latest therapy [e.g., radical surgery, transurethral resection of bladder tumor (TURBT), radiation, chemotherapy (neoadjuvant or adjuvant, or with radiation)]. Prior immune checkpoint inhibitor is not allowed.
      * Patient with history of >= pT4b, N+, and/or M1 UC is not eligible.
      * NOTE: Patients in whom concomitant or prior bladder/urethra predominant (>= 50%) urothelial carcinoma have been surgically resected and demonstrated to be only Ta or carcinoma in situ (CIS) (< cT1 N0) are eligible regardless of time elapsed
* Patient must not have any uncontrolled illness including, but not limited to, ongoing or active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), symptomatic congestive heart failure (CHF), myocardial infarction (MI) or unstable angina pectoris, significant uncontrolled cardiac arrhythmia, clinically relevant liver cirrhosis, interstitial lung disease, or psychiatric illness/social situations in the three months prior to registration that would limit compliance with study requirements
* Patient must not have received prior radiation therapy to >= 25% of the bone marrow for other diseases
* Patient must not have received prior systemic anthracycline therapy

  * NOTE: Patients who have received prior intravesical chemotherapy at any time for non-muscle invasive urothelial carcinoma of the bladder are eligible
* Patient must not have either history of or active autoimmune disease requiring immunosuppressive therapy within 2 years prior to registration/randomization or any history of inflammatory bowel disease (inflammatory bowel disease [IBD], e.g. ulcerative colitis, or Crohn's disease), neuromuscular autoimmune condition, immune-related pneumonitis or interstitial lung disease. Patients with well-controlled hyper/hypothyroidism, celiac controlled by diet alone, diabetes mellitus type I, vitiligo, alopecia, psoriasis, eczema, lichen planus, or similar skin/mucosa condition are eligible
* Patient must not be on or have used immunosuppressive medication within 14 days prior to the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, intra-auricular, topical steroids, or local steroid injections (e.g. intra-articular injection
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent at the time of enrollment
  * Steroids as pre-medications for hypersensitivity reactions (e.g. computed tomography [CT] pre-medication)
* Patient must not have received live attenuated vaccine within 30 days prior to the first dose of durvalumab, while on protocol treatment and within 30 days after the last dose of durvalumab
* Patient must not have had a major surgical procedure within 28 days prior to registration/randomization

  * NOTE: Cystoscopy/ureteroscopy, stent placement or nephrostomy tube is not considered major surgery
* Patient must not have history of allogenic organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) (Cisplatin eligible cohort: Arms A and B) | From registration/randomization to the earliest of systemic recurrence outside urinary tract, cancer progression, or death from any cause, assessed up to 5 years
  Disease progression prior to surgery or omission of surgery due to unresectable tumors, muscle-invasive cancer or disease recurring outside of the bladder, urethra, or contralateral upper tract are considered as events for EFS.
Pathologic complete response (pCR) (Cisplatin ineligible cohort: Arm C) | At surgery
  Will assess pathologic complete response at surgery (pCR, pT0N0/Nx) by local pathology review. Patients who drop out prior to surgery or who have unknown response status will be considered as non-responders.

SECONDARY OUTCOMES:
pCR (Cisplatin-eligible cohort: Arms A and B) | Up to 5 years
EFS (cisplatin-ineligible cohort: Arm C) | From registration/randomization to the earliest of systemic recurrence outside urinary tract, cancer progression, or death from any cause, assessed up to 5 years
  Will be characterized using the Kaplan-Meier method.
Overall survival (OS) (All Patients) | From registration/randomization to death from any cause, assessed up to 5 years
  OS will be evaluated by arm, post chemotherapy response (ypCR, stage yp =< T1N0, yp >= T2N0), as well as stage (ypCR and > ypCR) within and across treatment arms. Will be estimated using Kaplan-Meier method.
Urothelial cancer-free survival or disease-free survival (All Patients) | From the date of surgery to the earlier of a return of upper tract urothelial cancer (UTUC) or death from any cause, assessed up to 5 years
  A return of UTUC includes non-muscle invasive recurrences, pathologic T2 or higher muscle-invasive recurrences specifically in the urinary tract, metastatic disease outside the urinary tract, or death. Patients alive without documented UTUC will be censored at the date of last disease assessment.
Cancer-specific survival (All Patients) | From registration/randomization to death due to cancer; deaths due to other causes will be counted as competing events, assessed up to 5 years
  Will be analyzed using Gray's method and cumulative incidence estimates will be reported.
Renal function outcomes following systemic treatment and following radical nephroureterectomy (All Patients) | Post chemotherapy and post surgery
  The proportion of patients with renal insufficiency (creatinine [CrCl] < 60 ml/min) post chemotherapy and post nephroureterectomy as well as the proportion of patients with renal function improvement (CrCl < 60 ml/min at baseline and CrCl >= 60 ml/min on study) will be reported along with exact binomial confidence intervals. The distribution of changes in renal function post chemotherapy as well as post surgery from baseline will also be reported. The analysis of renal function outcomes will be performed among patients who receive at least one dose of study therapy.
Incidence of adverse events (All Patients) | Up to 30 days post surgery
  Toxicity will be evaluated in all treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean H Hoffman-Censits, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (257):
- United States (257):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm